CLINICAL TRIAL: NCT00932113
Title: An Investigator-Initiated, Assessor Blinded, Randomized Study Comparing the Mechanism of Action of Adalimumab to Methotrexate in Subjects With Moderate to Severe Chronic Plaque Psoriasis.
Brief Title: Mechanism of Action Study for Psoriasis
Acronym: MOA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MOA; ABT 08-030 (Other Grant/Funding Number: AbbVie)
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Psoriasis
Keywords: tumor necrosis factor (TNF) inhibitor; tumor necrosis factor (TNF) blockade; Methotrexate; treatment; mechanism; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate; Folic Acid; Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Active Comparator): Dosing will be on day 1 and then weekly. For the injections, dosing will occur according to product recommendations. Patients will receive 80mg adalimumab (2 pre-filled syringes, each with 40mg) on day 1, and then 40mg on week 1 and then every 2 weeks (from week 1 through week 15).
  Interventions: Drug: Adalimumab (Humira)
- Methotrexate (MTX) (Active Comparator): Patients will be dosed according to the CHAMPION study in single weekly doses of methotrexate: 7.5mg at week 0, 10mg at week two, and 15mg at week 4 for all patients. For each subject if the PASI did not decrease by at least 50% from baseline (PASI-50) at week 8, dosing will be increased to 20mg per week; the dose will be maintained at 15mg per week if PASI-50 was achieved at week 8. If PASI-50 was not achieved at week 12, dosing will be increased to 25mg per week; the dose will be maintained at 20mg per week if the PASI-50 was achieved at week 12. All patients on methotrexate will also receive a dietary supplement of oral folate (5mg per week). Methotrexate-treated patients will then receive 16 weeks of adalimumab at the end of study.
  Interventions: Drug: Methotrexate; Drug: Adalimumab (Humira)

INTERVENTIONS:
Drug: Methotrexate — 2 cohorts (Randomized 1:1 adalimumab:methotrexate). Subjects will receive treatment on Day 1 (baseline visit) and then weekly or every 2 weeks for 16 weeks.
  Methotrexate-treated patients will then receive 16 weeks of adalimumab at the end of study.
  Other Names: Methotrexate (MTX); Folic Acid
  Arms: Methotrexate (MTX)
Drug: Adalimumab (Humira) — 2 cohorts (Randomized 1:1 adalimumab:methotrexate). Subjects will receive treatment on Day 1 (baseline visit) and then weekly or every 2 weeks for 16 weeks.
  Other Names: Humira

SUMMARY:
The objective of this study is to compare the mechanism of action between adalimumab and methotrexate in subjects with psoriasis.

DETAILED DESCRIPTION:
Both methotrexate and adalimumab are FDA-approved drugs for the treatment of moderate to severe psoriasis. The two treatments, methotrexate and adalimumab, both show efficacy for psoriasis, however their profiles differ. In the CHAMPION Study, more adalimumab-treated, moderate to severe psoriasis patients achieved a PASI 75 after 16 weeks compared to those treated with methotrexate (80% vs. 36%). The reason for this difference is poorly understood. No direct comparative mechanism of action studies in psoriasis patients between methotrexate and adalimumab (or any tumor necrosis factor blocker) has been reported.

With etanercept, another tumor necrosis factor blocker, the in vivo mechanism has been studied with some scientific rigor. These studies demonstrate that etanercept down regulates multiple pro-inflammatory pathways (as shown in Table 1 of the protocol).

To date, there are no similar studies with adalimumab or methotrexate.

In order to understand the molecular and cellular basis for the differential clinical efficacy of adalimumab and methotrexate, it is essential to compare their mechanisms of action in psoriatic plaques. Biopsies will be performed, and we will study biomarkers in this proposal with immunohistochemistry, real-time polymerase chain reaction, and gene arrays.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-85 years of age with moderate to severe psoriasis, in general good health as determined by the PI based upon the results of medical history, laboratory profile, and physical examination, and who are candidates for systemic or phototherapy
* Presence of a psoriatic plaque of >2cm in an area which can be biopsied repeatedly.
* Men must agree to avoid impregnating a woman while on this study.
* Women are eligible to participate in the study if they meet one of the following criteria:

  * Women who are postmenopausal (>1 year), sterile, or hysterectomized
  * Women of childbearing potential must undergo monthly pregnancy testing during the study and agree to use two of the following methods of contraception throughout and for 60 days after the last dose of study drug:

    * Oral contraceptives
    * Transdermal contraceptives
    * Injectable or implantable methods
    * Intrauterine devices
    * Barrier methods (diaphragm or condom with spermicide)
    * Abstinence and Tubal Ligation are also considered a form of Birth control

Exclusion Criteria:

* Patients <18 or >85 years old
* Absence of a psoriatic plaque >2cm in diameter
* Active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit
* Evidence of skin conditions at screening (e.g. eczema) that would interfere with evaluations of the effect of study medication
* Inability to understand the consent process
* Receipt of any investigational drugs, psoralen+ultraviolet A or oral systemic treatments within 4 weeks of study drug initiation
* Biologics within 3 months of study initiation
* Topical steroids, topical vitamin A or D analog preparations, Ultraviolet B therapy or anthralin within 2 weeks of study drug initiation. (Exception-stable regimen of class I-II topical steroids on scalp, axillae, and groin)
* Methotrexate within 6 weeks of study initiation
* History of treatment with adalimumab
* History of primary non-response to methotrexate, infliximab or etanercept
* History of discontinuation of methotrexate or tumor necrosis factor (TNF) blocker for a safety-related reason that makes it unwise to restart either type of drug
* Any internal malignancy within 5 years (excluding fully excised cutaneous basal cell or squamous cell carcinoma)
* Pregnancy, not practicing effective birth control, or inability to practice safe sex during the length of the study
* Lactation
* Subjects who have known hypersensitivity to adalimumab or methotrexate or any of its components or who is known to have antibodies to etanercept
* History of alcohol or drug abuse one year before and during the study
* Known HIV-positive status or any other immune-suppressing disease
* Presence of a grade 3 or 4 infection <30 days prior to the screening visit, between the screening visit and the first day of treatment on study, or any time during the study that in the opinion of the PI would preclude participation in the study
* Any grade 3 or 4 adverse event, or laboratory toxicity, at the time of the screening visit or at any time during the study, which in the opinion of the PI would, preclude participation in the study

  * Serum creatinine >3.0 mg/dL (265 micromoles/L)
  * Serum potassium <3.5 mmol/L or > 5.5 mmol/L
  * Serum alanine aminotransferase or aspartate aminotransferase >3 times the upper limit of normal for the lab
  * Platelet count <100,000/mm3
  * White blood cell count <3,000/mm3
  * Hgb, Hct, or red blood cell outside 30% of the upper or lower limits of normal for the Lab
* Receipt of live vaccines 1 month prior to or while on study
* History of tuberculosis, and/or a positive PPD skin test/chest x-ray at screening without appropriate treatment-treatment of latent tuberculosis (for those with positive PPD tests) must be initiated prior to therapy with adalimumab or methotrexate
* Chronic hepatitis B or C infection, history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice B. Gottlieb, M.D., PhD., Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malaviya R, Sun Y, Tan JK, Magliocco M, Gottlieb AB. Induction of lesional and circulating leukocyte apoptosis by infliximab in a patient with moderate to severe psoriasis. J Drugs Dermatol. 2006 Oct;5(9):890-3. PMID 17039656
- [Background] Malaviya R, Sun Y, Tan JK, Wang A, Magliocco M, Yao M, Krueger JG, Gottlieb AB. Etanercept induces apoptosis of dermal dendritic cells in psoriatic plaques of responding patients. J Am Acad Dermatol. 2006 Oct;55(4):590-7. doi: 10.1016/j.jaad.2006.05.004. Epub 2006 Jul 3. PMID 17010737
- [Background] Gottlieb AB, Chamian F, Masud S, Cardinale I, Abello MV, Lowes MA, Chen F, Magliocco M, Krueger JG. TNF inhibition rapidly down-regulates multiple proinflammatory pathways in psoriasis plaques. J Immunol. 2005 Aug 15;175(4):2721-9. doi: 10.4049/jimmunol.175.4.2721. PMID 16081850
- [Background] Tan JK, Aphale A, Malaviya R, Sun Y, Gottlieb AB. Mechanisms of action of etanercept in psoriasis. J Investig Dermatol Symp Proc. 2007 May;12(1):38-45. doi: 10.1038/sj.jidsymp.5650037. PMID 17502868
- [Background] Lizzul PF, Aphale A, Malaviya R, Sun Y, Masud S, Dombrovskiy V, Gottlieb AB. Differential expression of phosphorylated NF-kappaB/RelA in normal and psoriatic epidermis and downregulation of NF-kappaB in response to treatment with etanercept. J Invest Dermatol. 2005 Jun;124(6):1275-83. doi: 10.1111/j.0022-202X.2005.23735.x. PMID 15955104
- [Result] Saurat JH, Stingl G, Dubertret L, Papp K, Langley RG, Ortonne JP, Unnebrink K, Kaul M, Camez A; CHAMPION Study Investigators. Efficacy and safety results from the randomized controlled comparative study of adalimumab vs. methotrexate vs. placebo in patients with psoriasis (CHAMPION). Br J Dermatol. 2008 Mar;158(3):558-66. doi: 10.1111/j.1365-2133.2007.08315.x. Epub 2007 Nov 28. PMID 18047523
- [Derived] Goldminz AM, Suarez-Farinas M, Wang AC, Dumont N, Krueger JG, Gottlieb AB. CCL20 and IL22 Messenger RNA Expression After Adalimumab vs Methotrexate Treatment of Psoriasis: A Randomized Clinical Trial. JAMA Dermatol. 2015 Aug;151(8):837-46. doi: 10.1001/jamadermatol.2015.0452. PMID 25946554

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The discrepancy between the enrollment number in the protocol section and number of participants in participant flow module is due to 3 participants screen failing and being allowed to re-screen. We counted them as enrolled upon signing of new consent and conducting re-screening visit.
Groups:
- Methotrexate (MTX): Patients dosed in single weekly doses of methotrexate 7.5mg at week 0, 10mg at week two, and 15mg at week 4 for all patients. For each subject if the PASI did not decrease by at least 50% from baseline (PASI-50) at week 8, dosing will be increased to 20mg per week; the dose will be maintained at 15mg per week if PASI-50 was achieved at week 8. If PASI-50 was not achieved at week 12, dosing will be increased to 25mg per week; the dose will be maintained at 20mg per week if the PASI-50 was achieved at week 12. All patients on methotrexate will also receive a dietary supplement of oral folate (5mg per week). Methotrexate-treated patients will then receive 16 weeks of adalimumab at the end of study.
  Methotrexate: 2 cohorts (Randomized 1:1 adalimumab:methotrexate). Subjects will receive treatment on Day 1 (baseline visit) and then weekly or every 2 weeks for 16 weeks.
  Methotrexate-treated patients will then receive 16 weeks of adalimumab at the end of study.
Period: Overall Study
Arm/Group | Adalimumab | Methotrexate (MTX)
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Methotrexate (MTX) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 50.5 [22 to 69] | 50.3 [22 to 69] | 50.4 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 11 | 13 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  caucasian | 12 | 14 | 26
  african american | 1 | 0 | 1
  unknown | 0 | 1 | 1
  hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Biologic Activity Endpoints
Description: Histologic and Immunohistochemistry endpoints; Relative messenger RNA gene expression (normalized to HARP); and Gene Arrays.
Time Frame: Weeks 0, 1, 2, 4 and 16
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Adalimumab | Methotrexate (MTX)
Number analyzed (Participants) | 15 | 15
fold change
  CAMP(responders) | -3.85 (0.79) | -2.83 (0.82)
  CAMP(Non responders) | 0.05 (2.2) | 0.84 (0.60)
  CCL20 (responders) | -3.55 (0.54) | -2.96 (0.51)
  CCL20 (non responders) | 0.84 (1.5) | 0.84 (0.6)
  CXCL1 (responders) | -3.01 (0.61) | -3.18 (0.7)
  CXCL1 (non responders) | 1.03 (1.6) | 1.22 (0.83)
  DEFB4A (responders) | -6.96 (0.96) | -6 (1.1)
  DEFB4A (non responders) | -0.07 (2.6) | 1.83 (1.2)
  IL 17F (responders) | -1.97 (0.99) | -3.24 (0.74)
  IL 17F (non responders) | 0.79 (2.8) | 1.02 (.87)
  IL 17A (responders) | -5.31 (0.98) | -4.75 (.96)
  IL 17A (non responders) | 0.18 (2.8) | 1.00 (1.1)
  IL 23 A (responders) | -3.90 (0.79) | -2.72 (0.56)
  IL 23A (non responders) | -0.81 (2.2) | 0.89 (0.67)
  IL 22 (responders) | -3.58 (1.0) | -5.14 (0.68)
  IL 22 (non rsponders) | 0.25 (2.8) | 1.00 (0.80)
  IFNG (responders) | -2.66 (0.77) | -1.77 (0.61)
  IFNG (non responders) | -0.52 (2.2) | 0.82 (0.72)
  MX1 (responders) | -1.90 (0.31) | -2.00 (0.46)
  MX1 (non responders) | 0.04 (0.86) | 0.47 (0.54)
Statistical Analysis 1: Comparison: Adalimumab vs Methotrexate (MTX); Test type: Other; p < 0.05, ANOVA

2. Secondary Outcome: Clinical Endpoints for Psoriasis: PASI 75
Description: PASI 75 is the percent of subjects who experience an improvement in PASI (Psoriasis Area and Severity Index) score of at least 75% from their baseline PASI score.
Time Frame: Weeks 0 and week 16
Measure: Number; unit: percentage of subjects
Arm/Group | Adalimumab | Methotrexate (MTX)
Number analyzed (Participants) | 15 | 15
percentage of subjects | 67 | 27

3. Other Pre Specified Outcome: Additional Gene Analysis (Ongoing)
Description: A single, long-term follow-up visit will be done for all available subjects for additional pharmacogenetic analysis. The goal in collecting DNA from psoriasis patients is to determine if individual subjects have gene variants associated with increased incidence of psoriasis. The investigators plan on analyzing variants using single nucleotide polymorphism (SNP) analysis by high-throughput DNA sequencing. This patient genetic information may allow us to correctly interpret data collected about gene expression levels in affected or non-affected skin. Additionally genetic typing may lead to cogent personalized health care (PHC) strategies for the identification of psoriasis drug responders/non-responders, patients who achieve durable disease remission post-treatment, and/or pharmacodynamic markers, as examples.
Time Frame: long-term follow-up visit 4- 6 years post end of study
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Endpoints for Psoriasis: Physician's Global Assessment (PGA) Clear or Almost Clear (PGA 0-1)
Time Frame: Week 0 and Week 16
Measure: Number; unit: percentage of subjects
Arm/Group | Adalimumab | Methotrexate (MTX)
Number analyzed (Participants) | 15 | 15
percentage of subjects | 73 | 27

5. Secondary Outcome: Clinical Endpoints for Psoriasis: % Body Surface Area
Time Frame: Week 0 and week 16
Measure: Mean (Full Range); unit: percentage of total body surface area
Arm/Group | Adalimumab | Methotrexate (MTX)
Number analyzed (Participants) | 15 | 15
percentage of total body surface area | 5.9 [0 to 25] | 10.7 [0 to 38]

6. Secondary Outcome: Clinical Endpoints for Psoriasis: Target Lesion Score
Description: The lesion score of a single psoriatic plaque selected at baseline. Total range is 0 - 12 with 0 being clear and 12 representing the most severe disease. The target lesion score is composed of scale, erythema, and induration, each parameter is scored 0 (clear) through 4 (very severe). Totals are summed for target lesion score. S+E+I = TLS
Time Frame: Week 0 and Week 16
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Adalimumab | Methotrexate (MTX)
Number analyzed (Participants) | 15 | 15
units on a scale | 1.2 [0 to 8.5] | 3.4 [0 to 9]

7. Secondary Outcome: Clinical Endpoints for Psoriasis: Photography Completed
Time Frame: Week 0 and Week 16
Measure: Number; unit: participants
Arm/Group | Adalimumab | Methotrexate (MTX)
Number analyzed (Participants) | 15 | 15
participants | 15 | 15

ADVERSE EVENTS:
Arm/Group | Adalimumab | Methotrexate (MTX)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=15) | Methotrexate (MTX) (N=15)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (5)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Biopsy Site Infection (Infections and infestations) | 1 (1) | 1 (1)
Flu-Like Symptoms (Infections and infestations) | 2 (2) | 1 (1)
Acute Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (10) | 6 (7)
Upper Respiratory Tract Infection/Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Epidermal Inclusion Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Biopsy of Nevi (Surgical and medical procedures) | 0 (0) | 1 (1)
Hair Loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Oral Apthous Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dislocated Thumb (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (Nervous system disorders) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Irritant Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Liquid Nitrogen to Skin Tag (Surgical and medical procedures) | 1 (1) | 0 (0)
Mood Swings (Psychiatric disorders) | 1 (1) | 0 (0)
Back Spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Injection Site Reaction/Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruise/abrasions s/p fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Finger Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ecchymoses near injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymoses near biopsy site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysesthesias (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No